CLINICAL TRIAL: NCT00061412
Title: Learning Disabilities: Links to Schools and Biology
Brief Title: Comprehensive Program to Improve Reading and Writing Skills in At-Risk and Dyslexic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2P50HD33812-6; 2P50HD033812 (NIH)
Record Dates: First submitted 2003-05-27; First posted 2003-05-28 (Estimated); Last update posted 2006-09-28 (Estimated); Status verified 2006-09

CONDITIONS: Dyslexia; Learning Disorders
Keywords: Low reading and writing achievement; At-risk students; Reading Disability; Writing Disability
MeSH Terms: conditions — Dyslexia; Learning Disabilities

INTERVENTIONS:
Behavioral: Comprehensive program to improve reading and writing skills

SUMMARY:
This project is evaluating programs to improve reading and writing skills in children who have or are at risk for having reading disabilities. The project focuses on children who are at-risk for low achievement in school and on children with dyslexia.

DETAILED DESCRIPTION:
This study is part of a larger project to investigate the biological and educational constraints operating in children with learning disabilities, with a focus on treatment and links between assessment and treatment. The project evaluates prevention and treatment of reading and writing disabilities, the genetic contribution to subtypes of dyslexia, the relationship between brain variables and dyslexia, and the brain's response to treatment for dyslexia. Genetic and brain imaging studies occur throughout the project.

During Year 1, at-risk readers in first grade were targeted for an intervention for mapping spoken words onto written words. These students were compared to a control group. During Year 2, the faster responders (those who reached grade level) and the slower responders (those who were not yet at grade level) from Year 1 were compared. Slower responders received additional treatment and comparisons were made again at the end of the year. The additional treatment was also studied in Spanish-speaking students in first grade. During Year 3, another group of at-risk, poor readers in second grade were randomized to either word decoding treatment, comprehension treatment, a combined word decoding and comprehension treatment, or a control treatment.

During Year 4, readers at risk for failing state standards in reading (decoding) participated in an extended day program providing comprehensive reading instruction. The students were compared to a control group. During Year 5, all students grades 4 to 9 took a battery of morphological, reading, and writing tests. The testing was administered throughout an entire school system.

During Year 6, older students with dyslexia were randomly assigned to phonological or morphological reading training. Students were then compared on pre- and post-test behavioral measures and brain activation results. During Year 7, students with dyslexia were randomly assigned to an orthographic or morphological treatment for spelling. Students underwent brain imaging before and after the intervention. Behavioral and brain activation measures were also assessed. During Year 8, students with dyslexia underwent attention or fluency training and writing training with and without attentional bridges. Only behavioral measures were collected.

Recruitment of families for the family genetics study is ongoing. Recruitment for the brain imaging-treatment studies will begin in 2004 when installation of new brain imaging equipment is complete.

ELIGIBILITY:
Inclusion Criteria

* Student in grades 1 to 9
* Underachieving in reading and writing
* English as first language

Exclusion Criteria

* Mental retardation
* Developmental disability such as autism or pervasive developmental disorder
* Brain damage or disease affecting brain function
* Severe language or psychiatric disorder

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500
Dates: Start 1995-12; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Berninger, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Eckert MA, Leonard CM, Richards TL, Aylward EH, Thomson J, Berninger VW. Anatomical correlates of dyslexia: frontal and cerebellar findings. Brain. 2003 Feb;126(Pt 2):482-94. doi: 10.1093/brain/awg026. PMID 12538414
- [Background] Richards TL, Berninger VW, Aylward EH, Richards AL, Thomson JB, Nagy WE, Carlisle JF, Dager SR, Abbott RD. Reproducibility of proton MR spectroscopic imaging (PEPSI): comparison of dyslexic and normal-reading children and effects of treatment on brain lactate levels during language tasks. AJNR Am J Neuroradiol. 2002 Nov-Dec;23(10):1678-85. PMID 12427623
- [Background] Hsu L, Wijsman EM, Berninger VW, Thomson JB, Raskind WH. Familial aggregation of dyslexia phenotypes. II: paired correlated measures. Am J Med Genet. 2002 May 8;114(4):471-8. doi: 10.1002/ajmg.10523. PMID 11992573
- [Background] Corina DP, Richards TL, Serafini S, Richards AL, Steury K, Abbott RD, Echelard DR, Maravilla KR, Berninger VW. fMRI auditory language differences between dyslexic and able reading children. Neuroreport. 2001 May 8;12(6):1195-201. doi: 10.1097/00001756-200105080-00029. PMID 11338191
- [Background] Berninger VW, Abbott RD, Brooksher R, Lemos Z, Ogier S, Zook D, Mostafapour E. A connectionist approach to making the predictability of English orthography explicit to at-risk beginning readers: evidence for alternative, effective strategies. Dev Neuropsychol. 2000;17(2):241-71. doi: 10.1207/S15326942DN1702_06. PMID 10955205
- See also: Click here for more information on this trial. — http://depts.washington.edu/coe/programs/ep/profiles/faculty/berninger.html